CLINICAL TRIAL: NCT02782221
Title: Lipolytic Effects of GH in Human Subjects in Vivo: Molecular Mechanisms and Temporal Patterns
Brief Title: Lipolytic Effects of GH in Human Subjects in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GH02
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Diseases; Growth Hormone Treatment
Keywords: lipolysis; ATGL
MeSH Terms: conditions — Metabolic Diseases | interventions — Growth Hormone; Human Growth Hormone; pegvisomant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth hormone (Active Comparator): Subjects are receiving growth hormone
  Interventions: Drug: Growth Hormone
- Placebo (Placebo Comparator): Subjects are receiving pegvisomant to block the action of growth hormone
  Interventions: Drug: Pegisomant

INTERVENTIONS:
Drug: Growth Hormone — Subjects are receiving one injection of growth hormone (Genotropin) 0,5 mg
  Other Names: Genotropin
  Arms: Growth hormone
Drug: Pegisomant — One the placebo day the subjects are receiving injection with pegvisomant (Somavert 30 mg) to block the action of endogenous growth hormone
  Other Names: Somavert
  Arms: Placebo

SUMMARY:
Growth hormone (GH) induces fat metabolism. The mechanisms underlying the fat metabolizing effects of GH remain elusive. However, it is known that insulin suppresses fat metabolism, and GH inhibits the expression of certain insulin-dependent signaling proteins. We therefore hypothesize that the fat metabolizing effects of GH depend on abrogation of insulin-dependent signaling pathways.

In order to investigate the fat metabolizing effects of GH, we'll analyze consecutive adipose tissue biopsies taken after GH exposure and GH blocking, respectively.

Knowledge of the effects of growth hormone and fat metabolism can in shot-sight as well as in long-sight have great importance for the understanding of growth disorders from overweight and type 2 diabetes to malnutrition and eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* no medication
* BMI 28-35

Exclusion Criteria:

* known diseases
* regular medication

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Lipolytic activity measured as area under the curve (AUC) for FFA (blood sample). | 1 year

SECONDARY OUTCOMES:
Substrate metabolism as measured by indirect calorimetry | 3 months
GH signaling proteins in adipose tissue measured by western blotting | 1,5 years
Intracellular lipolytic activity measured by an ATGL assay | 1 year
GH signaling gene targets in adipose tissue measured by qPCR | 1,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator — University Hospital of Aarhus
Locations (1):
- University Hospital of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nielsen TS, Jessen N, Jorgensen JO, Moller N, Lund S. Dissecting adipose tissue lipolysis: molecular regulation and implications for metabolic disease. J Mol Endocrinol. 2014 Jun;52(3):R199-222. doi: 10.1530/JME-13-0277. Epub 2014 Feb 27. PMID 24577718
- [Background] Moller N, Jorgensen JO. Effects of growth hormone on glucose, lipid, and protein metabolism in human subjects. Endocr Rev. 2009 Apr;30(2):152-77. doi: 10.1210/er.2008-0027. Epub 2009 Feb 24. PMID 19240267
- [Derived] Hjelholt AJ, Lee KY, Arlien-Soborg MC, Pedersen SB, Kopchick JJ, Puri V, Jessen N, Jorgensen JOL. Temporal patterns of lipolytic regulators in adipose tissue after acute growth hormone exposure in human subjects: A randomized controlled crossover trial. Mol Metab. 2019 Nov;29:65-75. doi: 10.1016/j.molmet.2019.08.013. Epub 2019 Aug 20. PMID 31668393